CLINICAL TRIAL: NCT00391105
Title: Comparative Study of the Use of Remifentanil Versus Morphine for Sedation and Analgesia of Premature Neonates During Mechanical Ventilation in the Treatment of Respiratory Distress Syndrome (RDS)
Brief Title: Remifentanil Versus Morphine for Sedation of Premature Neonates With Respiratory Distress Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ETIC 287/04
Record Dates: First submitted 2006-10-19; First posted 2006-10-23 (Estimated); Last update posted 2006-10-23 (Estimated); Status verified 2006-10

CONDITIONS: Respiratory Distress Syndrome
Keywords: intubation; Sedation; Analgesia; preterm neonate; remifentanil; morphine; respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome; Agnosia | interventions — Remifentanil

INTERVENTIONS:
Drug: Remifentanil

SUMMARY:
In this randomised controlled study we intended to compared intubation conditions and the continuous infusion of remifentanil (n=10) and morphine (n=10) in mechanically ventilated premature neonates (28-34wk) regarding the time to be awake and, the time until extubation after interruption of the opioid administration.

DETAILED DESCRIPTION:
Intubation and mechanical ventilation are majors component of intensive care for premature neonates with respiratory distress syndrome (RDS) and is associated with physiologic, biochemical, and clinical responses indicating pain and stress in prematures. Although morphine is one of the most used drugs for premedication and for sedation and analgesia during mechanical ventilation in the treatment of RDS its pharmacological profile precludes several limitations mostly due to its much delayed onset of action what makes the drug not suitable as premedication and due to its prolonged duration of action mainly in prematures. Unlike morphine, remifentanil has an unique pharmacokinetic properties with a rapid onset of action and, a fast decrease in plasma concentration after interruption of administration due to a context-sensitive half-time of 3.2 minutes. So, it could be the ideal opioid for neonates who are especially sensitive to respiratory depression by opioids

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 28 and 34 wk
* Clinical and radiological features compatible with respiratory distress syndrome that required an elective tracheal intubation and surfactant therapy.

Exclusion criteria:

* The presence of major congenital malformations
* Birth weigh less than 1000g
* Previous or concurrent use of opioid for any reason (cesarean section with general anaesthesia)
* Hemodynamic instability before the indication of tracheal intubation
* Refuse of the parents to enroll the neonate in the study protocol

Ages: 60 Minutes to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2004-04; Study Completion 2005-11

PRIMARY OUTCOMES:
Intubation conditions using a four point scale
Decrease in time after interruption of sedation until the neonate be awake.
Decrease in time after interruption of sedation until the neonate be extubated.

SECONDARY OUTCOMES:
Pain and stress before and after intubation (NIPS and Comfort scores).
Pain and stress during continuous infusion of remifentanil versus morphine during mechanical ventilation for the treatment of respiratory distress syndrome (NIPS and Comfort scores).

CONTACTS AND LOCATIONS:
Overall Officials: Yerkes P Silva, MD, MSc, Principal Investigator — Faculty of Medicine from Federal University of Minas Gerais

REFERENCES:
- [Background] Pereira e Silva Y, Gomez RS, Barbosa RF, Simoes e Silva AC. Remifentanil for sedation and analgesia in a preterm neonate with respiratory distress syndrome. Paediatr Anaesth. 2005 Nov;15(11):993-6. doi: 10.1111/j.1460-9592.2005.01666.x. PMID 16238563